CLINICAL TRIAL: NCT00169286
Title: Organized Self-management Support for Chronic Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: R21MH065530 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression

INTERVENTIONS:
Procedure: Telephone care management
Procedure: peer-led chronic disease self-management workshop
Procedure: professionally-led cognitive behavioral psychotherapy group

SUMMARY:
This study aims to adapt and pilot test two core elements of an organized care program (systematic telephone outreach and monitoring to improve quality and continuity of pharmacotherapy, and structured psychoeducational group programs focused on patient activation and self-management) in a population-based sample of patients with chronic or recurrent depression.

DETAILED DESCRIPTION:
This study aims to adapt and pilot test two core elements of an organized care program (systematic telephone outreach and monitoring to improve quality and continuity of pharmacotherapy, and structured psychoeducational group programs focused on patient activation and self-management) in a population-based sample of patients with chronic or recurrent depression. Two forms of group self-management training will be evaluated: a Peer-Led Chronic Disease Self-Management Group (after that developed by Lorig and colleagues) and a Therapist-Led Cognitive-Behavioral Therapy Group. Approximately 100 patients with chronic or recurrent depression were randomly assigned to one of four conditions: 1) usual care; 2) phone care management; 3) phone care management plus peer-led self-management group; or 4) phone care management plus therapist-led CBT group. Blinded assessments will examine clinical outcomes (SCL depression score, depression diagnosis by SCID), functional outcomes, and process variables (self-efficacy for managing depression, use of coping strategies) over 12 months. If patients choose not to participate in treatment, reasons for dropout were assessed. The data collected will provide:1) an evaluation of the feasibility and acceptability (including recruitment, intervention uptake and continued participation) of the intervention programs; 2) preliminary evaluation of effectiveness, i.e., the effects of each intervention on patient outcomes and process of care; and 3) information to inform the design and implementation of a full-scale effectiveness trial (refinement of intervention programs and measurement strategy, necessary sample size).

ELIGIBILITY:
Inclusion Criteria:

* history of at least one major depression in the last two years
* history of recurent major depression or dysthymia
* significant residual symptoms after 6 months of treatment

Exclusion Criteria:

* history of mania or hypomania
* cognitive impairment
* near-terminal medical illness
* intent to disenroll from health plan

emergent clinical needs

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104
Dates: Start 2003-07; Study Completion 2005-06

PRIMARY OUTCOMES:
feasibility and acceptability (including recruitment, intervention uptake and continued participation) of the intervention programs

SECONDARY OUTCOMES:
clinical outcomes (SCL depression score, depression diagnosis by SCID), functional outcomes (SF-36 Questionnaire, and process variables (self-efficacy for managing depression)

CONTACTS AND LOCATIONS:
Overall Officials: Evette J Ludman, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States